CLINICAL TRIAL: NCT02121288
Title: A Randomized, Open-Label, Parallel, Multi-Center, Phase IV Study to Assess the Effect of Ticagrelor vs Clopidogrel on Adenosine-Induced Myocardial Blood Flow in Peripheral Artery Disease (PAD)Patients
Brief Title: Adenosine-induced Myocardial Blood Flow in Peripheral Artery Disease Patients
Acronym: PAD
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D5135L00001
Record Dates: First submitted 2014-04-22; First posted 2014-04-23 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Peripheral Artery Disease; Vascular Disease; Arterial Occlusion Disease; Intermittent Claudication; Ankle Brachial Index (0.9 or Less)
Keywords: Peripheral Artery Disease; Myocardial Blood Flow; Cardiac Blood Flow
MeSH Terms: conditions — Peripheral Arterial Disease; Vascular Diseases; Intermittent Claudication | interventions — Ticagrelor; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ticagrelor (Experimental): oral ticagrelor 90 mg (yellow) tablet
  Interventions: Drug: Ticagrelor
- Clopidogrel (Active Comparator): oral clopidogrel 75 mg (pink) tablet
  Interventions: Drug: clopidogrel

INTERVENTIONS:
Drug: Ticagrelor — Day 1: Loading dose of ticagrelor 180mg (two 90mg tablets) followed by 90mg dose at 12 hours after loading dose. Subject continues to take ticagrelor 90mg twice a day (morning and evening) for 7 days until next visit (Day 7).
  Other Names: Brilinta
  Arms: Ticagrelor
Drug: clopidogrel — Day 1: Clopidogrel 75mg oral tablet. Subjects will continue to take clopidogrel 75mg once a day for 7 days until next visit (Day 7/Visit 3). Note: no loading dose is given for the clopidogrel as those subjects are already on chronic dosing.
  Other Names: Plavix
  Arms: Clopidogrel

SUMMARY:
The purpose of the study is to assess the effect of blood flow to the heart when subjects are treated with ticagrelor (Brilinta) or clopidogrel (antiplatelet drugs that stop the blood from clumping together) in patients with Peripheral Artery Disease (PAD).

DETAILED DESCRIPTION:
The effects of ticagrelor and clopidogrel on adenosine-induced myocardial blood flow (MBF) will be evaluated by cardiac 13N- ammonia positron emission tomography (PET) at rest (baseline), acute dosing on Day 1, and at short term dosing on Day 7.

Subjects receiving ticagrelor will have additional pharmacokinetic (PK) blood samples collected at specific time points to measure ticagrelor concentration in the blood. Subjects' participation will be approximatetly 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic lower extremity PAD defined by:
* Symptoms at the time of screening including classic claudication, other exertional leg discomfort associated with physical limitations from PAD, AND Ankle brachial index (ABI) measurement at Visit 1 needs to be < 0.90. OR, Prior lower extremity revascularization for symptomatic and haemodynamically significant PAD greater than 30 days prior to randomisation, irrespective of present leg symptoms and the Ankle Brachial Index (ABI).
* Male and female ≥ 18 years of age and less than 60 yrs.
* Subjects must be taking clopidogrel (75mg/day) for at least 30 days prior to entry to study.

Exclusion Criteria:

* Participation in another clinical study with an investigational product during the last 30 days.
* History of ACS within the last 1 year.
* Hypersensitivity or contraindications to clopidogrel or ticagrelor.
* Need for chronic oral anticoagulant therapy or chronic low- molecular-weight heparin or long-term treatment with fondaparinux, warfarin, apixaban, rivoroxaban, and parenteral anticoagulants such as enoxeparin, and bivalirudin.
* Life expectancy < 6 months based on investigator's judgment.
* Planned lower extremity revascularization (surgical or endovascular) in any vascular territory within the next 3 months or with current ischemic ulcers or gangrene.
* Planned major amputation due to PAD within the next 3 months or major amputation due to PAD within the last 30 days.
* Subjects who have suffered a stroke during the past 3 months.
* Dementia likely to jeopardize understanding of information pertinent to study conduct or compliance to study procedures
* Severe hypertension that may put the subject at risk.
* Subjects considered to be at risk of bradycardic events (e.g., known sick sinus syndrome or second or third degree AV block unless already treated with a permanent pacemaker.
* Known severe liver disease (e.g., ascites and/or clinical signs of coagulopathy).
* Renal failure requiring dialysis
* A known bleeding diathesis, haemostatic or coagulation disorder, or systemic bleeding, whether resolved or ongoing
* History of previous intracranial bleed at any time, gastrointestinal bleed within the past 6 months, or major surgery within 30 days (if the surgical wound is judged to be associated with an increased risk of bleeding).
* History of thrombocytopenia or neutropenia
* Females of child-bearing potential (i.e., those who are not chemically or surgically sterilized, post-menopausal who are not willing to use an accepted method of treatment OR who have a positive pregnancy test at screening.
* Concern for inability of the subject to comply with study procedures and/or follow-up (e.g., alcohol or drug abuse).

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2014-12; Primary Completion 2016-02 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Assessment of ticagrelor when compared to clopidogrel on adenosine-induced myocardial blood flow (MBF) by cardiac 13N ammonia Positron EmissionTomography (PET) at Visit 2 | Visit 2 (Day 1): 1 day treament visit
  Assess the acute treatment effects on the 13N-ammonia PET measure and evaulate if they can be correlated with plasma exposure of ticagrelor and or its active metabolite. Subjects will recieve 180mg ticagrelor loading dose or no loading dose for clopidogrel arm, since those subjects are already on chronic dosing. Subjects will undergo additional adenosine-PET at 2 hours following ticagrelor or 4 hours following clopidogrel administration to ascertain MBF.

SECONDARY OUTCOMES:
Assessment of ticagrelor when compared to clopidogrel on adenosine-induced myocardial blood flow (MBF) by cardiac 13N ammonia Positron EmissionTomography (PET) at Vist 3 | Visit 3 (Day 7): occurs 7 days after Visit 2
  Assess the short-term treatment effects on the 13N-ammonia PET measure and evaulate if they can be correlated with plasma exposure of ticagrelor and or its active metabolite. The same sequence described at Visit 2 will be repeated during Visit 3.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Budoff, MD, Principal Investigator — Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center; Gabriel Vorobiof, MD, Principal Investigator — University of California, Los Angeles